CLINICAL TRIAL: NCT06034561
Title: Bortezomib-based Regimen for Refractory or Relapsed Acute Lymphoblastic Leukemia in Adults
Brief Title: Bortezomib-based Regimen for Refractory or Relapsed Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4009/23
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia With Failed Remission
Keywords: Acute lymphoblastic leukemia; Bortezomib; Salvage therapy; Bridge therapy; Response rate
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib; Vincristine; Doxorubicin; pegaspargase; Dexamethasone; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib (Experimental): Patients with refractory or relapsed acute lymphoblastic leukemia will receive one-two courses of salvage regimen composed by:
  * Bortezomib 1.3 mg/m2 I.V. D1,D4,D8,D11;
  * Vincristine 1.5 mg/m2 I.V. (maximum at 2 mg) - D1, D8,D15,D22;
  * Doxorubicin 60 mg/m2 I.V. - D1;
  * Peg-asparaginase 2000 IU/m2 I.V. - D4 and D18;
  * Dexamethasone 20 mg/m2 P.O. or I.V. (divided BID) - D1-D5 and D15-D19
  * Intrathecal chemotherapy: methotrexate 12 mg + dexamethasone 2 mg.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Patients should receive one or two courses of this regimen, aiming to achieve complete remission as a bridge to proceed with allogeneic HSCT.
  Other Names: Vincristine; Doxorubicin; Peg-asparaginase; Dexamethasone; Methotrexate

SUMMARY:
This is a interventional phase II study aiming to examine the complete response rate of a bortezomib-based salvage regimen in adults with refractory or relapsed acute lymphoblastic leukemia (ALL), seeking to compare outcomes with the available literature and with our historical data on relapsed/refractory ALL.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is a rare neoplasm in adults, with long-term survival rates approaching 50% with current regimens. Although high rates of complete response are achieved with the first-line therapy, many patients are primary refractory or may further relapse. Arguably, these patients have a more resistant disease with higher risk genetic alterations and a much less likely to be cured, which almost always only can be obtained by a following allogeneic hematopoietic stem-cell transplantation (HSCT). Therefore, strategies to salvage patients with detectable disease after induction blocks or with relapsed disease are crucial to prolong survival and potentially cure those patients, working as a bridge therapy to HSCT. Historically, patients with relapsed/refractory ALL have received multidrug regimens based on high-dose cytarabine, such as fludarabine, cytarabine and idarubicin (FLAG-IDA). Those regimens provide a 30-40% complete response rate with non-negligible toxicity. Recently, new targeted agents such as blinatumomab, inotuzumab, and cellular therapies have arisen for B-lineage disease, even though these agents are not available in the public health setting. Previous studies have tested salvage regimens for ALL encompassing proteasome inhibitors plus highly synergistic drugs (dexamethasone, vincristine, asparaginase, doxorubicin), with exciting outcomes in limited case series. For adults, these regimens are less studied. However, preliminary data suggest that they are less toxic and more potent since patients can receive different drug combinations that they had not been exposed to before. The primary objective of this study is to examine the complete response rate of this regimen in our population, aiming to compare with the available literature and with our historical data on relapsed/refractory ALL. Secondary objectives are:

1. To determine the safety and feasibility of a bortezomib-based regimen for salvage relapsed/refractory ALL in our setting.
2. To determine the rate of patients who are able to proceed with HSCT after the treatment.
3. To calculate event-free survival and overall survival after the salvage regimen for relapsed/refractory ALL.
4. To calculate the rate of measurable residual disease (MRD) negative status after the treatment.
5. To examine the rate of febrile neutropenia, liver toxicity, neurotoxicity, and treatment-related mortality after this regimen in relapsed/refractory ALL.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 16 and 60 years-old with refractory or relapsed ALL (≥1% of anomalous blasts by flow cytometry in bone marrow or peripheral blood) after one or two lines of therapy, regardless of their phenotype or baseline genetic alteration;
* Patients are eligible after allogeneic HSCT as long as patients are not actively being treated for graft-versus-host-disease (GvHD).

Exclusion Criteria:

* Burkitt leukemia;
* Prior myeloproliferative disease;
* Drug allergies;
* Eastern Cooperative Oncology Group (ECOG) scale >2;
* Total bilirubin>2x upper limit of normal (ULN);
* Transaminases>5x ULN;
* Creatinine>2,5 mg/dl;
* Active uncontrolled infection;
* History of asparaginase-induced pancreatitis;
* Prior exposure to bortezomib;
* Heart failure New York Heart Association (NYHA) Class III or IV;
* Patients with more than 400mg/m2 lifetime exposure of anthracycline;
* Severe psychiatric disorder which prevents adequate compliance;
* Refusal to participate in the study.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Complete response | 30 days
  Disappearance of lymphoid blasts in peripheral blood, with fewer than 5% of lymphoid blasts quantified in the bone marrow aspirate through immunophenotyping.

SECONDARY OUTCOMES:
Event-free survival | 1 year
  Time interval between study enrollment and the occurrence of an event (non-response, relapse, or death) or last follow-up (censorship).
Overall survival | 1 year
  Time interval between study enrollment and the occurrence of death or last follow-up (censorship).
Rate of MRD-negativity | 60 days
  Absence of pathological lymphoid blasts in a bone marrow sample detected through immunophenotyping with a minimum sensitivity of 10-4.
Rate of allogeneic hematopoietic stem-cell transplantation | 1 year
  Proportion of patients who successfully underwent allogeneic hematopoietic stem-cell transplantation after the study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Wellington Silva, MD PhD, Principal Investigator — Instituto do Cancer do Estado de Sao Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No